CLINICAL TRIAL: NCT06376955
Title: High Intensity Interval Exercise Versus Focused Ultrasound on Insulin Resistance in Diabetic Female Patients With Abdominal Obesity
Brief Title: High Intensity Interval Versus Focused Ultrasound on Insulin Resistance in Diabetics With Abdominal Obesity
Acronym: diabetic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Fouad Abd-Elrahman, Departments of physical therapy for women's health, Faculty of Physical Therapy, Badr University in Cairo., Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-1
Record Dates: First submitted 2024-04-16; First posted 2024-04-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Insulin Resistance; Abdominal Obesity; Diabetes
MeSH Terms: conditions — Insulin Resistance; Obesity, Abdominal; Diabetes Mellitus | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A High intrerval trainig exercise group (Experimental): Group A will receive high intensity interval exercise 2 times per week for 4 months in addition to intermitted fasting diet.
  Interventions: Other: High intensity interval exercise
- Group B Focused ultrasound group (Experimental): Group B will receive focused ultrasound 2 times per week for 4 months in addition to intermitted fasting diet.
  Interventions: Other: Focused ultrasound

INTERVENTIONS:
Other: High intensity interval exercise — HIIT is a type of interval training exercise. It incorporates several rounds that alternate between several minutes of high intensity movements followed by short periods of lower intensity movements 2 times per week for 4 months.
  Arms: Group A High intrerval trainig exercise group
Other: Focused ultrasound — Focused ultrasound will be applied over the anterior abdominal, two sessions per week for 4 months, each session 40 minutes.
  Arms: Group B Focused ultrasound group

SUMMARY:
Obesity and diabetes share a common insulin resistance pathway and contribute to chronic hyperglycemia. Both high-intensity interval exercise (HIIE) and focused ultrasound (FUS) have been explored in the context of managing insulin resistance in diabetic individuals with abdominal obesity, though they operate through different mechanisms and have different implications.

DETAILED DESCRIPTION:
Forty diabetic females aged 25 to 35 years old and body mass index was ≥ 30 kg/m², will participate in this study. They will be assigned into two equal groups, Group A will receive high intensity interval exercise 2 times per week for 4 months in addition to intermitted fasting diet. Group B will receive focused ultrasound 2 times per week for 4 months in addition to intermitted fasting diet. Assessment of abdominal obesity will be applied pre and post treatment through measuring Body mass index (BMI), Waist circumference (WC) in addition to Value of HbA1c and HOMA-IR hormone will be measured to determine effect of treatment on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

They will be recruited from El_shinnawy physical therapy Centre.

* All are suffering from abdominal obesity
* Their age between 25-35 years old
* Their body mass index more than 30 kg/m2,
* Their waist circumference ranged from 88 cm
* The fat thickness at the treatment area was at least 2.5 cm

Exclusion Criteria:

* Females having any skin diseases in the abdomen.
* Female suffering from any physical or mental disorders.
* Females suffering from abdominal scars or hernia
* Females didn´t take any medication that might affect their weight all over the study period.
* Females complaining from any cardiovascular disorders.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-08 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Body mass index | Before starting the study and after 4 months of treatment
  The weight and height of each woman in both groups will be measured to calculate the body mass index (BMI)
Waist circumference | Before starting the study and after 4 months of treatment
  Assessment of waist circumference of each woman by the tape measurement
Skin fold | Before starting the study and after 4 months of treatment
  The thickness of the abdominal fold will be measured using skinfold calipers to provide information on changes in subcutaneous fat in the abdominal region.
Value of HbA1c and HOMA-IR hormone | Before starting the study and after 4 months of treatment
  Value of HbA1c and HOMA-IR hormone will be measured to determine effect of treatment on insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Elshinnawy, Assistant, Principal Investigator — Horus University; Haitham M. Elmasry, Lecturer, Principal Investigator — MTI University; Shimaa hussien ahmed roshdy, Lecturer, Principal Investigator — Misr University for Science and Technology